CLINICAL TRIAL: NCT01625845
Title: Targeting Systemic Inflammation to Concurrently Treat Late-Life Depression and Reduce Coronary Artery Disease Risk
Brief Title: Anti-INFLammatory to Address Mood and Endothelial Dysfunction (INFLAMED)
Acronym: INFLAMED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1110007119; R24MH080827 (NIH); 1737 (Other: Indiana Clinical Research Center)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-10

CONDITIONS: Major Depressive Disorder; Depression; Depressive Symptoms; Cardiovascular Disease (CVD); Coronary Artery Disease (CAD); Heart Disease
Keywords: Major Depressive Disorder; Depression; Depressive Symptoms; Cardiovascular Disease (CVD); Coronary Artery Disease (CAD); Heart Disease; Endothelial Function; Inflammation
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Cardiovascular Diseases; Coronary Artery Disease; Heart Diseases; Inflammation | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pentoxifylline + Standard Treatment (Experimental): Pentoxifylline: Pentoxifylline is phosphodiesterase inhibitor that interferes with proinflammatory cytokine signaling and synthesis. Participants will be instructed to take pentoxifylline 400 mg p.o. t.i.d. for 12 weeks.
  Standard Treatment: Beating the Blues (BtB) is a widely used, empirically supported, computer-based, CBT program for depression designed for use in primary care clinics. BtB utilizes an interactive, multimedia format to deliver and eight 50-minute, weekly therapy sessions.
  Interventions: Drug: Pentoxifylline; Behavioral: Standard Treatment
- Placebo + Standard Treatment (Placebo Comparator): Placebos: Placebo pills will match the study drug for color, taste, texture, size, and smell. Participants will receive the same instructions as those randomized to pentoxifylline.
  Standard Treatment: Beating the Blues (BtB) is a widely used, empirically supported, computer-based, CBT program for depression designed for use in primary care clinics. BtB utilizes an interactive, multimedia format to deliver and eight 50-minute, weekly therapy sessions.
  Interventions: Other: Placebo; Behavioral: Standard Treatment

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline 400 mg p.o. t.i.d. for 12 weeks
  Other Names: Trental; Pentoxil; Pentopak
  Arms: Pentoxifylline + Standard Treatment
Other: Placebo — Placebo pills will match the study drug for color, taste, texture, size, and smell. Participants will receive the same instructions as those randomized to pentoxifylline.
  Arms: Placebo + Standard Treatment
Behavioral: Standard Treatment — BtB is a widely used, empirically supported, computer-based, CBT program for depression designed for use in primary care clinics. BtB utilizes an interactive, multimedia format to deliver and eight 50-minute, weekly therapy sessions. General topics covered include identifying and challenging automatic thoughts, cognitive errors, core beliefs, and attributional styles; activity scheduling; problem solving; graded exposure; task breakdown; sleep management; and relapse prevention. In addition to session work, patients are assigned homeworks that are customized to their needs and reviewed at the start of each session. A progress report, including whether the patient is experiencing suicidal ideation, is generated at the end of each session.
  Other Names: Computer-Based Cognitive Behavioral Therapy (CBT); Computer-Based Psychotherapy

SUMMARY:
The objective of this clinical trial is to evaluate whether an anti-inflammatory medication, pentoxifylline, reduces depressive symptoms and improves artery function. Participants in this trial will be older primary care patients (60 years and up) who are depressed but do not have a history of cardiovascular disease. Half of these patients will receive pentoxifylline, and half will receive placebo. In addition, participants in both arms will receive an evidence-based psychological treatment called Beating the Blues®, which is a computerized, cognitive behavioral treatment program for depression. The investigators will use questionnaires to assess change in depressive symptoms and an ultrasound test to measure change in artery function from pre- to post-treatment. It is hypothesized that patients who receive pentoxifylline will show greater improvements in both depression and artery function than patients who receive placebo.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death, and depression is the leading cause of disability in the United States. Previous research suggests that systemic inflammation may play an important role in the development of both depression and cardiovascular disease. Therefore, Aim #1 of this study is to examine whether adding an anti-inflammatory medication (pentoxifylline) to standard depression treatment (cognitive-behavioral therapy) improves both depressive symptoms and endothelial dysfunction, a sign of early cardiovascular disease. Aim #2 is to evaluate candidate mediators of treatment effects by examining whether reductions in multiple markers of systemic inflammation account for treatment-related improvements in depressive symptoms and endothelial dysfunction. To achieve these aims, a clinical trial of older depressed primary care patients free of cardiovascular disease is being conducted. Patients will be randomized to one of two groups: a standard depression treatment (a cognitive-behavioral treatment program) plus pentoxifylline or standard depression treatment plus placebo. The treatment phase of the study will be 12 weeks. At baseline, 6 weeks, and 12 weeks, patients will undergo assessments of depressive symptoms, various inflammatory markers, and endothelial function. Our index of endothelial function is brachial artery flow-mediated dilation, a noninvasive measure of endothelial function. Demonstrating that medications targeting systemic inflammation are effective for concurrently treating late-life depression and reducing CAD risk would place anti-inflammatory approaches in the collection of depression treatment strategies, as well as CAD prevention strategies, of the primary care provider. This change to clinical practice should result in improved management of both late-life depression and cardiovascular risk, which in turn would reduce disability, CAD morbidity, and mortality among older adults.

ELIGIBILITY:
Inclusion Criteria:

* Primary care patients
* Age ≥ 40 years
* Clinically significant depressive symptoms, defined as a PHQ-9 score ≥15
* English speaking

Exclusion Criteria:

* History of clinical cardiovascular disease
* History of cardiac arrhythmias or cardiomyopathy
* History of carotid bruits
* History of certain chronic disorders (HIV/AIDS, kidney disease, liver disease, systemic inflammatory disease, or past-year cancer)
* History of bleeding disorder, gastrointestinal ulceration or bleeding, cerebrovascular aneurysm or bleeding, or retinal hemorrhage
* History of migraine headaches
* History of Raynaud's phenomenon
* History of bipolar disorder or psychosis
* Current use of anticoagulants or vasodilators (Lipid-lowering antihypertensive medications are allowed.)
* Current use of acetazolamide, anticonvulsants, or thyroid replacements
* Current use of glucocorticoids - including topical, nasal, or oral steroids - or anabolic steroids (Physiologic testosterone replacement therapy is allowed.)
* Current use of anti-inflammatory agents (including, but not limited to, plaquenil, infliximab, etanercept, mycophenolate mofetil, sirolimus, tacrolimus, cyclosporine, pentoxifylline, thalidomide)
* Known allergy or intolerance to pentoxifylline or other methylxanthines, such as , theophylline, caffeine, theobromine
* Known allergy or intolerance to nitroglycerin.
* Severe cognitive impairment (≥3 errors on 6-item cognitive screen105)
* Current alcohol use problem (≥2 on CAGE questionnaire106)
* Very severe depressive symptoms, defined as a PHQ-9 score ≥24
* Acute risk of suicide
* Vision or hearing problems
* Unable to lie flat for 30 minutes at a time
* Therapy for acute infection or other serious medical illnesses within 14 days prior to the pre-treatment visit (Therapy for acute infection or other serious medical illnesses that overlaps with a main study visit will result in postponement of that study visit until the course of therapy is completed; postponement outside of the allowed study visit timeframe will result in study discontinuation.)
* Creatinine clearance < 50mL/min using a serum creatinine level measured at the pre-treatment visit
* Hemoglobin < 9.0mg/dL at the pre-treatment visit
* Alanine aminotransferase (ALT) level or aspartate aminotransferase (AST) > 3 times ULN at the pre-treatment visit
* Total bilirubin > 2.5 times ULN at the pre-treatment visit
* Current evidence of abuse of prescription medications
* Current evidence of illicit drug use

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse C Stewart, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University-Purdue University Indianapolis (IUPUI), Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was open from June 28, 2012 to February 28, 2014. Participants were recruited from Eskenazi Health and Indiana University Health primary care clinics in Indianapolis. 1369 patients were screened, of whom 36 (2.6%) were eligible and provided informed consent. 16 patients (44%) attended the pre-treatment visit and were randomized.
Period: Overall Study
Arm/Group | Pentoxifylline + Standard Treatment | Placebo + Standard Treatment
Started | 10 | 6
Completed | 5 | 3
Not Completed | 5 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pentoxifylline + Standard Treatment | Placebo + Standard Treatment | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Brachial Flow-Mediated Dilation (FMD) From Pre- to Post- Treatment
Description: Patients underwent ultrasound assessment of brachial FMD in accordance with established guidelines at pre- (0 weeks) and post- (12 weeks) treatment. After a 10-minute supine rest, high-resolution baseline images of the brachial artery were obtained from 3 consecutive cardiac cycles. Next, the forearm cuff was inflated to 250 mmHg for 5 minutes and then was rapidly deflated. At 60 and 90 seconds post-deflation, images from 3 consecutive cardiac cycles were acquired. FMD values were computed as the % change in brachial diameter at either 60 or 90 seconds after cuff deflation
Time Frame: 0 and 12 weeks
Measure: Mean (Standard Error); unit: % change in brachial diameter
Arm/Group | Pentoxifylline + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 5 | 3
% change in brachial diameter | -1.18 (1.48) | 0.79 (1.95)
Statistical Analysis 1: Comparison: Pentoxifylline + Standard Treatment vs Placebo + Standard Treatment; Test type: Superiority or Other; p = .474, ANCOVA

2. Primary Outcome: Change in Depressive Symptoms Severity (Hopkins Symptom Checklist Depression Scale; SCL-20) From Pre- to Post- Treatment
Description: Self-reported depressive symptom severity was measured at pre- (0 weeks) and post- (12 weeks) treatment visits by the 20 depression items from the Symptom Checklist 90 (Hopkins Symptom Checklist depression scale; SCL-20). Each item on the scale ranges from 0 (not at all) to 4 (extremely). Total scores are the average across all response items and range from 0 to 4 with higher scores indicating greater levels of depressive symptoms.
Time Frame: 0 and 12 weeks
Measure: Mean (Standard Error); unit: Change in Total Score
Arm/Group | Pentoxifylline + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 5 | 3
Change in Total Score | -0.35 (0.25) | -1.41 (0.34)
Statistical Analysis 1: Comparison: Pentoxifylline + Standard Treatment vs Placebo + Standard Treatment; Test type: Superiority or Other; p = .068, ANCOVA

3. Secondary Outcome: Change in Circulating Tumor Necrosis Factor-Alpha (TNF-a) From Pre- to Post-Treatment
Description: A marker of systemic inflammation measured from blood samples collected at pre- and post-treatment.
Time Frame: 0 and12 weeks
Population: Participants with missing TNF-a data were excluded from this analysis.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Pentoxifylline + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 3 | 2
pg/mL | -0.65 (0.08) | -0.47 (0.10)
Statistical Analysis 1: Comparison: Pentoxifylline + Standard Treatment vs Placebo + Standard Treatment; Test type: Superiority or Other; p = .296, ANCOVA

4. Secondary Outcome: Change in Circulating Interleukin-6 (IL-6) From Pre- to Post-Treatment
Description: A marker of systemic inflammation measured from blood samples collected at pre- and post-treatment.
Time Frame: 0 and 12 weeks
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Pentoxifylline + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 5 | 3
pg/mL | -0.69 (1.02) | 1.84 (1.34)
Statistical Analysis 1: Comparison: Pentoxifylline + Standard Treatment vs Placebo + Standard Treatment; Test type: Superiority or Other; p = .203, ANCOVA

5. Secondary Outcome: Change in Circulating Interleukin-10 (IL-10) From Pre- to Post-Treatment
Description: An anti-inflammatory cytokine measured from blood samples collected at pre- and post-treatment.
Time Frame: 0 and 12 weeks
Population: One participant, with extreme outlier values at pre- and post-treatment, was excluded from analyses.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Pentoxifylline + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 5 | 2
pg/mL | -0.58 (0.34) | -0.66 (0.54)
Statistical Analysis 1: Comparison: Pentoxifylline + Standard Treatment vs Placebo + Standard Treatment; Test type: Superiority or Other; p = .906, ANCOVA

6. Secondary Outcome: Change in Interleukin-1ra (IL-1ra) From Pre- to Post-Treatment
Description: A marker of systemic inflammation measured from blood samples collected at pre- and post-treatment.
Time Frame: 0 and 12 weeks
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Pentoxifylline + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 5 | 3
pg/mL | 2.32 (75.03) | 25.00 (99.55)
Statistical Analysis 1: Comparison: Pentoxifylline + Standard Treatment vs Placebo + Standard Treatment; Test type: Superiority or Other; p = .869, ANCOVA

7. Secondary Outcome: Change in Circulating C-Reactive Protein (CRP) From Pre- to Post-Treatment
Description: A marker of systemic inflammation measured from blood samples collected at pre- and post-treatment.
Time Frame: 0 and 12 weeks
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Pentoxifylline + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 5 | 3
mg/L | -0.49 (1.34) | 6.44 (1.74)
Statistical Analysis 1: Comparison: Pentoxifylline + Standard Treatment vs Placebo + Standard Treatment; Test type: Superiority or Other; p = .026, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse event data were collected the recruitment initiation in June 2012 until study completion in May 2014. For each participant, adverse event data were collected between the pre- and post-treatment visits.
Description: A brief questionnaire created by the investigators was administered at each study visit to identify potential adverse events. Each event was evaluated by the study physician, who also provided severity and study involvement ratings. Clinical management decisions were made by the study physician in conjunction with the participant's provider(s).
Arm/Group | Pentoxifylline + Standard Treatment | Placebo + Standard Treatment
Serious Adverse Events (participants affected / at risk) | 3/10 | 0/6
Other Adverse Events (participants affected / at risk) | 8/10 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentoxifylline + Standard Treatment (N=10) | Placebo + Standard Treatment (N=6)
Complications after removing nodules during endoscopy (Chest pain, esophagitis, dizziness, bleeding) (General disorders) | 1 (1) | 0 (0)
Nasolabial abscess (Facial swelling) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hearing issues after explosion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentoxifylline + Standard Treatment (N=10) | Placebo + Standard Treatment (N=6)
Hemolyzed blood sample (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Flushed (General disorders) | 1 (1) | 2 (2)
Hot flashes (General disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 3 (3) | 3 (3)
Facial Pimple (General disorders) | 0 (0) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leg swelling (General disorders) | 0 (0) | 1 (1)
Headaches (General disorders) | 3 (3) | 0 (0)
Abnormalities in the complete blood cell count (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heartburn (General disorders) | 1 (1) | 0 (0)
Racing heart (General disorders) | 1 (1) | 0 (0)
Red eye (General disorders) | 1 (1) | 0 (0)
Diarrhea (General disorders) | 3 (3) | 0 (0)
Blurred vision (General disorders) | 2 (2) | 1 (1)
Impaired fasting glucose (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Low energy (General disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Sleep disturbance (General disorders) | 1 (1) | 0 (0)
Stomach Pain (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nervousness / jittery hands (General disorders) | 1 (1) | 0 (0)
Leg pain (General disorders) | 1 (1) | 0 (0)
Back pain (General disorders) | 1 (1) | 0 (0)
Sweating (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Missing data precluded analysis of two secondary outcome variables: IL-1α and IL-1β.

Due to the very small sample of randomized patients, conclusions should not be drawn from the results of this pilot trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No